CLINICAL TRIAL: NCT05440812
Title: Evaluation of the Effectiveness of a Newly Developed Blended Module for Patients Recovering from Depression (STAIRS): a Mixed Methods Randomized Controlled Trial
Brief Title: Improving Personal Recovery After Depression with a Blended Module (STAIRS)
Acronym: STAIRS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Hanze University of Applied Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202100347
Record Dates: First submitted 2022-06-21; First posted 2022-07-01 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Depression
Keywords: personal recovery
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Efficacy of STAIRS will be assessed by conducting a randomized controlled trial (N=140). In this trial, participants will be randomly assigned either to the experimental group receiving care as usual complemented with the STAIRS-training or the control group receiving care as usual. Measurement points are at T0 (baseline), T1 (post-treatment) and T2 (6 months after end of treatment). Qualitative semi-structured interviews will be held in the experimental group at T1 about the value that participants assign to the elements of the training, as well as the experienced acceptability, and perceived usefulness of the training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care As Usual plus STAIRS (Experimental): Care as usual added with a eight week STAIRS-training
  Interventions: Behavioral: Storytelling and Training to Advance Individual Recovery Skills (STAIRS)
- Care As Usual (No Intervention): Care as usual added with three information letters

INTERVENTIONS:
Behavioral: Storytelling and Training to Advance Individual Recovery Skills (STAIRS) — STAIRS is a 8-week program, in which 8 different themes are addressed. Coverage of each theme starts with a group meeting guided by a professional and expert by experience. In these meetings different exercises are done (e.g., filling out an actual and desired week-schedule, role-playing a difficult situation), information is given and experiences are shared. Between meetings, participants can choose from a range of homework exercises to practice their desired skills in a tailored way. In addition, participants can share experiences with the other group members and exchange reactions using a private online community.
  Arms: Care As Usual plus STAIRS

SUMMARY:
Almost all mental healthcare treatments of depression focus on symptomatic recovery. However, such recovery does not inherently mean that personal recovery is reached. In fact, many persons still experience functional impairments after symptomatic recovery. As this has a negative influence on daily life, a new blended module (STAIRS) was developed to promote personal recovery in persons that are in the final stage of symptomatic recovery from depression. The current study will investigate the efficacy of STAIRS, by adding STAIRS to care as usual and comparing it with care as usual. It is hypothesized that STAIRS will have a positive effect on personal recovery and that this effect is larger than in the control group.

DETAILED DESCRIPTION:
The study uses a mixed methods design to determine efficacy and underlying mechanisms contributing to the effect of the STAIRS-training. One hundred forty adults, who are in the last phase of their depression treatment, will be enrolled and randomized (1:1) to (1) a group receiving the STAIRS-training next to Care as Usual (CAU) or (2) a group receiving CAU added with three information letters. Level of personal recovery, symptom severity, empowerment and control will be determined at baseline, at the end of the program (8 weeks) and at 6 months follow up. Approximately fifteen participants from the STAIRS group will be asked about their experiences with the different elements of the program and the perceived effects, in a semi-structured interview at the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old
* Being in the last phase (recovery phase) of treatment for a diagnosed Major Depressive Disorder; psychological treatment is expected to end within three months or treatment is finished within the past 3 months and patient receives an aftercare and/or maintenance antidepressant treatment.
* No more than moderate depression severity: Score of <38 on the Inventory of Depressive Symptomatology - Self Rated (IDS-SR).
* The willingness to participate: an affirmative response to the question 'after being explained what participation means for you, are you willing to participate?'.

Exclusion Criteria:

* Bipolar depression or depression with psychotic features.
* Comorbid schizophrenia spectrum or other psychotic disorder.
* Comorbid moderate or severe dependence of alcohol or drugs.
* Neurological disorder (e.g., dementia).
* Insufficient command of the Dutch language.
* Cognitive problems or indication of low IQ (i.e.< 80).
* Not in possession of a pc or smartphone.
* Having been referred to a different mental health service for other mental problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Inventory Recovery Outcome Counter (I.ROC) total score | Baseline, end of treatment (8 weeks) and 6 months follow up
  The I.ROC is a self report rating scale containing 12 items measuring the level of personal recovery. Each item is rated on a 6-point ordinal scale, ranging from 0 (never) to 5 (always). Total scores range from 0 to 72. A higher score is better.
Change from baseline in Recovery Assessment Scale, Domains and Stages (RAS-DS) total score | Baseline, end of treatment (8 week) and 6 months follow up
  The RAS-DS is a self report rating scale containing 38 items measuring the level of personal recovery. Each item is rated on a 4-point ordinal scale, ranging from 0 (untrue) to 4 (completely true). Total scores range from 0 to 152. A higher score is better.

SECONDARY OUTCOMES:
Change from baseline in Inventory of Depressive Symptomatology - Self Report (IDS-SR) total score | Baseline, end of treatment (8 weeks) and 6 months follow up
  The IDS-SR is a self report rating scale containing 30 items, of which 28 need to be answered, measuring the level of depressive symptom severity. Each item is rated on a 4-point ordinal scale, ranging from 0 to 3. Total scores range from 0 to 84. A higher score is worse.
Change from baseline in Sheehan Disability Scale (SDS) total score | Baseline, end of treatment (8 week) and 6 months follow up
  The SDS is a self report rating scale containing 5 items, measuring the level of global functional impairments caused by symptoms. Three items are rated on a 11-point ordinal scale, ranging from 0 (not at all) to 10 (extremely). Total scores range from 0 to 30. A higher score is worse. Furthermore two items measure the number of days lost or unproductive caused by symptoms.
Depression relapse in the last six months, diagnosed with the Dutch version of the Mini International Neuropsychiatric Interview - Simplified (M.I.N.I - S), section MDEp | 6 months follow up
  The Dutch version of the M.I.N.I. (MINI-S voor DSM-5 Nederlandse versie 2019, Overbeek & Schruers / English - Version 2 © Hergueta & Weiller, 2017) is a structured diagnostic interview for diagnosing psychiatric disorders. Section MDEp is used to diagnose the presence or absence of DSM-5 Major Depressive Disorder (MDD) in the past six months.
Change from baseline in Netherlands Empowerment List (NEL) total score | Baseline, end of treatment (8 weeks) and 6 months follow up
  The NEL is a self report rating scale containing 40 items measuring the level of empowerment. Each item is rated on a 5-point ordinal scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Total scores range from 40 to 200. A higher score is better.
Change from baseline in Mastery Scale total score | Baseline, end of treatment (8 weeks) and 6 months follow up
  The Mastery Scale is a self report rating scale containing 7 items measuring the level of control over events and ongoing situations. Each item is rated on a 5-point ordinal scale, ranging from 0 (strongly disagree) to 4 (strongly agree). Total scores range from 0 to 28. A higher score is better.
Change from baseline in Self-Management Ability Scale (SMAS-30) total score | Baseline, end of treatment (week 8) and 6 months follow up
  The SMAS-30 is a self report rating scale containing 30 items measuring the level of self-management. Each item is rated on a 6-point ordinal scale, ranging from 1 to 6. Total scores range from 30 to 180. A higher score is better.
Economic evaluation, based on the Treatment Inventory of Costs in Psychiatric patients | Baseline, end of treatment (8 weeks) and 6 months follow up
  The TIC-P is a self report questionnaire measuring the medical costs and productivity losses caused by health problems related to psychiatric disorders.
Perceived effects and program valuation by patients recovering from a depression | End of intervention (8 weeks)
  User experiences on program elements considered helpful, investigated with a semi structured interview with selected participants from the STAIRS-group containing questions about what helped them in which way in their personal recovery process
Acceptability and usability of the STAIRS-training for patients recovering from a depression | End of intervention (8 weeks)
  User experiences on acceptability and usability, investigated with a semi structured interview containing questions about the content, didactics and organization of the meetings, homework assignments and used website.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Schoevers, prof, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - GGZ Drenthe, Assen, Drenthe
  - University Medical Center Groningen, Groningen, Provincie Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wedema D, Wardenaar KJ, Alma MA, van Asselt ADI, Korevaar EL, Schoevers RA. A blended module (STAIRS) to promote functional and personal recovery in patients with a major depressive disorder in remission: study protocol of a concurrent mixed methods randomized controlled trial. BMC Psychiatry. 2023 Oct 7;23(1):727. doi: 10.1186/s12888-023-05213-w. PMID 37805486
- See also: official website of the intervention — http://stairstraining.nl